CLINICAL TRIAL: NCT04762212
Title: Examining the Effects of a Posterolateral Mobilization With Movement (MWM) and a Dynamic Stretch With Over Pressure on Hip Flexion: A Randomized Control Trial.
Brief Title: Examining the Effects of a Mobilization With Movement and a Dynamic Stretch With Over Pressure on Hip Flexion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Cathy Arnot, Clinical Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00103113
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Hip; Anomaly
MeSH Terms: conditions — Congenital Abnormalities | interventions — Movement

STUDY DESIGN:
Intervention Model Description: A parallel design, also called a parallel group study, compares two or more treatments. Participants are randomly assigned to either group, treatments are administered, and then results are compared.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The care provider (Cathy Arnot) will not be blinded as she knew the groups of the participants. The Investigators and the Outcomes Assessors were blinded as they were not aware of the group each participant was placed in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip with the greatest limitation in flexion range of motion (Active Comparator): Participants that have limited hip flexion of less than 101 degrees will be randomly assigned to one of two groups: one intervention group will receive Mobilization with Movement and home program of stretching with over-pressure one group will receive only a home program of stretching with over-pressure.
  Interventions: Procedure: Mobilization with movement and stretching, stretching or control
- Hip with the least limitation in flexion range of motion (Active Comparator): Participants least limited hip in flexion range of motion will serve as the control group. This limb will not receive an intervention.
  Interventions: Procedure: Mobilization with movement and stretching, stretching or control

INTERVENTIONS:
Procedure: Mobilization with movement and stretching, stretching or control — The participants will receive a therapist performed mobilization with movement and then instructed in a stretching program to be followed for one week or only receive instruction in a stretching program to be followed for one week on the hip with the greatest limitation in motion. The hip with the least amount of limitation will not receive an intervention.

SUMMARY:
The purpose of this study is to compare the effects of a mobilization with movement (MWM) technique performed by a physical therapist with those of a dynamic stretch with over pressure on active hip flexion range of motion (ROM) in those with active hip flexion ROM limitations. There is limited evidence available in the literature examining the therapeutic effects of MWM at the hip, the long term effects of MWM, or whether one modality is more effective than another. This study seeks to address these gaps in the literature by directly comparing the results of these two manual therapy interventions on active hip flexion ROM.

DETAILED DESCRIPTION:
This study aims to compare the effects of a therapist-performed mobilization with movement (MWM) technique with those of a dynamic stretch with over pressure on active hip flexion range of motion (ROM) in those with active hip flexion ROM limitations.Those individuals from the University of South Carolina's Department of Physical Therapy (UofSC DPT) community who are interested in becoming study participants will be identified by means of announcements made in the Seminar in Physical Therapy course which is attended by all students, faculty, and staff of UofSC DPT each week. Interested individuals will be provided with Cathy Arnot's email address in order to schedule an evaluation session to determine whether or not they meet the study's inclusion and exclusion criteria. In addition, Sarah Cooper will attend a staff meeting at Vertex PT Specialists to make an announcement and provide the attendees with Cathy Arnot's email for inquiries. Participants will be assigned to either the MWM group or the dynamic stretch with over pressure group via blocked randomization for sex and age, with at least seventeen participants being placed into each group. The MWM group participants will receive a therapist-performed MWM technique and a prescription for a home exercise program (HEP) consisting of a dynamic stretch with over pressure to be performed once a day over the course of the following week. The dynamic stretch with over pressure group participants will receive only the prescription for the HEP consisting of the dynamic stretch with over pressure to be performed once a day over the following week. Measurements will be assessed at four time points: Immediately before the intervention, immediately after the intervention, 24 hours after the intervention, and one week after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The sole inclusion criterion will be a limitation in hip flexion to less than 101 degrees in both hips.

Exclusion Criteria:

* Any traumatic injury to or surgical procedure performed upon the lower extremities within the last six months
* Any contraindication to dynamic stretching, weight-bearing rotation, or MWM of the hip joint
* Any dermatologic pathology in the area of the strap application
* Any pain provoked by active hip flexion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Degrees of change in hip flexion range of motion will be measured using a goniometer at baseline. | Baseline
  Degrees of hip flexion range of motion will be measured before intervention with the participant in supine .All measurements will be taken using a goniometer which measures range of motion in degrees from 0-360.
Degrees of change in hip flexion range of motion will be measured using a goniometer immediately after intervention. | Immediately post-intervention.
  Degrees of hip flexion range of motion will be measured immediately after intervention with the participant in supine .All measurements will be taken using a goniometer which measures range of motion in degrees from 0-360.
Degrees of change in hip flexion range of motion will be measured using a goniometer 24 hours after intervention. | 24 hours after intervention.
  Degrees of hip flexion range of motion will be measured 24 hours after intervention with the participant in supine. All measurements will be taken using a goniometer which measures range of motion in degrees from 0-360.
Degrees of change in hip flexion range of motion will be measured using a goniometer one week after intervention. | 1 week after intervention.
  Degrees of hip flexion range of motion will be measured one week after intervention with the participant in supine. All measurements will be taken using a goniometer which measures range of motion in degrees from 0-360.
Star Excursion Balance Test (SEBT) at baseline | Baseline.
  The participants will perform the posterior, posterolateral, and posteromedial portions of the SEBT. The SEBT is standardized test the participant stands in the center of a mat with "stars" in 8 directions. The particpant stands on one foot and reaches with their opposite foot as far as they can without losing balance. It is method to measure functional hip flexion.
Star Excursion Balance Test (SEBT) immediately post-intervention | Immediately post-intervention.
  The participants will perform the posterior, posterolateral, and posteromedial portions of the SEBT. The SEBT is standardized test the participant stands in the center of a mat with "stars" in 8 directions. The particpant stands on one foot and reaches with their opposite foot as far as they can without losing balance. It is method to measure functional hip flexion.
Star Excursion Balance Test (SEBT) 24 hours after intervention | 24 hours after intervention.
  The participants will perform the posterior, posterolateral, and posteromedial portions of the SEBT. The SEBT is standardized test the participant stands in the center of a mat with "stars" in 8 directions. The particpant stands on one foot and reaches with their opposite foot as far as they can without losing balance. It is method to measure functional hip flexion.
Star Excursion Balance Test (SEBT) one week after intervention | 1 week after intervention.
  The participants will perform the posterior, posterolateral, and posteromedial portions of the SEBT. The SEBT is standardized test the participant stands in the center of a mat with "stars" in 8 directions. The particpant stands on one foot and reaches with their opposite foot as far as they can without losing balance. It is method to measure functional hip flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy F Arnot, DPT, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No